CLINICAL TRIAL: NCT00905177
Title: Predictors of Anticoagulation Control on Warfarin Therapy
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 700902
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Heart Valve Replacement
Keywords: Atrial Fibrillation; deep vein thrombosis; anticoagulation; warfarin; coumadin
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A one time blood sample will be collected for specific genetic testing and vitamin K assay
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this research study is to develop better dosing of anticoagulation medication in both Caucasian and African Americans through analysis of various genetic factors.

DETAILED DESCRIPTION:
This is a prospective cohort study among adult patients requiring warfarin therapy. Patients presenting for anticoagulation will be identified at the start of therapy and followed throughout their course until they reach maintenance dose. We will then develop a dosing equation for warfarin using patient, environmental and genetic factors.

ELIGIBILITY:
Inclusion Criteria:

* All Caucasians and African Americans who are new to warfarin therapy

Exclusion Criteria:

* Under 21 years of age
* Non caucasian
* Non african american
* Have an abnormal INR before warfarin or heparin therapy
* Unable to provide consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include all self-identified Caucasians and African Americans initiating warfarin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 687 (Actual)
Dates: Start 2009-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E. Kimmel, M.D. MS, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Anticoagulation Management Center, Philadelphia, Pennsylvania
  - Philadelphia Veteran Affairs Medical Center, Philadelphia, Pennsylvania